CLINICAL TRIAL: NCT04658745
Title: Effects of Theta Burst Stimulation on Modulation of Mirror Illusion-induced Rhythm Suppression in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20171106002-01
Record Dates: First submitted 2020-11-30; First posted 2020-12-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Hemiplegia
Keywords: Stroke; upper extremity; intermittent theta burst stimulation; mirror visual feedback; event-related desynchronization
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iTBS over the ipsilesional primary motor cortex plus mirror therapy (Experimental): iTBS: iTBS (20 trains of ten bursts at eight-second intervals, 600 stimuli, 200-second per session) will be delivered to the ipsilesional hemisphere in stroke patients. After the iTBS therapy, participants will practice the movements with the non-affected hand and try moving the affected arm at the same time to synchronize with the non-affected hand (illusion on the mirror). The movement practice will involve 5 table-top tasks and the participant will be instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session, lasting for 20 minutes.
  Interventions: Device: Intermittent theta burst stimulation; Behavioral: Mirror Therapy
- Sham iTBS over the ipsilesional primary motor cortex plus mirror therapy (Sham Comparator): iTBS (20 trains of ten bursts at eight-second intervals, 600 stimuli, 200-second per session) will be delivered to the ipsilesional hemisphere, but with a sham coil (i.e., sham iTBS). After the sham stimulation, participants will practice the movements with the non-affected hand and try moving the affected arm at the same time to synchronize with the non-affected hand (illusion on the mirror). The movement practice will involve 5 table-top tasks and the participant will be instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session, lasting for 20 minutes.
  Interventions: Behavioral: Mirror Therapy; Device: Sham intermittent theta burst stimulation
- iTBS to the ipsilesional primary motor cortex plus sham mirror therapy (Sham Comparator): iTBS (20 trains of ten bursts at eight-second intervals, 600 stimuli, 200-second per session) will be delivered to the ipsilesional hemisphere in stroke patients. After the iTBS therapy, participants will practice the movements with the non-affected hand and try moving the affected arm at the same time, but with a covered mirror (e.g., sham mirror therapy).
  In the sham mirror therapy condition, the mirror is covered by a cloth and the participant is instructed to move both arms while looking at a cross mark on the covered mirror and imaging the analogous movements of the affected arm. The movement practice will involve 5 table-top tasks (same as mirror therapy) and the participant will be instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session, lasting for 20 minutes.
  Interventions: Device: Intermittent theta burst stimulation; Behavioral: Sham mirror Therapy

INTERVENTIONS:
Device: Intermittent theta burst stimulation — iTBS (20 trains of ten bursts at eight-second intervals, 600 stimuli, 200-second per session) will be delivered to the ipsilesional hemisphere in stroke patients, by using a butterfly shape coil.
  Arms: iTBS over the ipsilesional primary motor cortex plus mirror therapy; iTBS to the ipsilesional primary motor cortex plus sham mirror therapy
Behavioral: Mirror Therapy — Participants will practice the movements with the non-affected hand and try moving the affected arm at the same time to synchronize with the non-affected hand (illusion on the mirror). The movement practice will involve 5 table-top tasks and the participant will be instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session, lasting for 20 minutes.
  Arms: Sham iTBS over the ipsilesional primary motor cortex plus mirror therapy; iTBS over the ipsilesional primary motor cortex plus mirror therapy
Device: Sham intermittent theta burst stimulation — iTBS (20 trains of ten bursts at eight-second intervals, 600 stimuli, 200-second per session) will be delivered to the ipsilesional hemisphere in stroke patients. However, a sham coil will be used, which is not associated with any stimulation effect on the brain.
  Arms: Sham iTBS over the ipsilesional primary motor cortex plus mirror therapy
Behavioral: Sham mirror Therapy — In sham mirror therapy, the mirror will be covered. Participants will practice the movements with the non-affected hand and try moving the affected arm at the same time to move the non-affected hand. The participants cannot receive mirror visual feedback of the paretic upper extremity movement during the therapy. Same as mirror therapy, the movement practice will involve 5 table-top tasks and the participant will be instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session, lasting for 20 minutes.
  Arms: iTBS to the ipsilesional primary motor cortex plus sham mirror therapy

SUMMARY:
The study aims to test the hypothesis that rTMS in the form of theta burst stimulation (TBS) over the ipsilateral and contralateral motor cortices can modulate mirror illusion-induced rhythm suppression while observing unilateral arm movement in stroke individuals. The investigators further hypothesize that this intervention will lead to the revision of interhemispheric asymmetry. Finally, this study will also explore the longitudinal relationship between rhythm suppression and motor recovery as indicated by motor excitability in the form of MEP. The results of this study will provide significant new information regarding neurophysiological motor relearning mechanisms which could inform the development and evaluation of innovative treatments for individuals with stroke

DETAILED DESCRIPTION:
Stroke is the leading cause of physical disability. Facilitating the process of motor relearning would greatly accelerate the rehabilitation of motor functions and elicit positive neuroplasticity of the damaged brain area. Previous research has already explored the feasibility of motor priming techniques embedded in stroke rehabilitation programs using strategies such as non-invasive brain stimulation (NIBS) and mirror therapy (MT). These treatments are usually implemented along with the standardized rehabilitation, sequentially or simultaneously, and have been demonstrated to be more effective than the standardized rehabilitation programs alone.

Mirror neuron, as indicated traditionally by the decrease in the amplitude of Mu rhythm, i.e. a suppression over central electrodes of electroencephalography (EEG), reflects the "seeing" of movement after "perception". Such oscillations are based on neural substrates that are discharged during the observation and execution of a motor act, which is also associated with other human functions, such as imitation, language, etc. The core mirror neuron system (MNS) is thought to be located in the premotor and the primary sensorimotor cortices, indicating that motor learning could be enhanced during action observation and overt movement.

Preliminary research has shown that repetitive Transcranial Magnetic Stimulation (rTMS) can enhance the corticomotor excitability in mirror neurons during both observation of movement (by others) or imagined movement in healthy subjects; in particular, as measured by enhanced motor evoked potentials (MEP). Increases in MEP has also been induced by short-term action observation and mirror visual feedback in stroke survivors. However, it is not yet known if MNS can be activated by TMS in MT following a stroke, and the relationship between mirror neuron activation and clinical improvements in stroke remains unclear.

The investigators have already published preliminary findings in patients with hemiplegic upper extremity, rTMS, and MT. Here, the investigators propose to test the hypothesis that rTMS in the form of theta-burst stimulation (TBS) over the ipsilateral and contralateral motor cortices can modulate mirror illusion-induced rhythm suppression while observing unilateral arm movement in stroke individuals. The investigators further hypothesize that this intervention will lead to the revision of interhemispheric asymmetry. Finally, this study will also explore the longitudinal relationship between rhythm suppression and motor recovery as indicated by motor excitability in the form of MEP. The results of this study will provide significant new information regarding neurophysiological motor relearning mechanisms which could inform the development and evaluation of innovative treatments for individuals with stroke

ELIGIBILITY:
Inclusion Criteria:

1. type and location of stroke - ischemic or hemorrhagic, cortical or subcortical, confirmed by medical diagnoses compatible with a unilateral lesion involvement;
2. Acute stroke patients: stroke with onset of neurological condition ≤3 months, recruited from a local hospital; Chronic stroke patients: stroke with onset of neurological condition from 6 months to 3 years, recruited from self-help organization in the community. The randomization will be pre-stratified into 2 - subacute and chronic stages, and recruit from 2 centers - acute hospital and self-help organizations in the community.
3. normal or corrected-to-normal visual acuity better than 20/60 (6/18) in the better eye;
4. right-handed, verified by the Edinburgh Handedness Inventory;
5. mild to moderately impaired hemiplegic upper extremity functions, with functional levels 5-7 as rated by the Functional Test for the Hemiplegic Upper Extremity - Hong Kong version (FTHUE-HK);
6. the ability to understand and follow simple verbal instructions;
7. the ability to participate in a therapy session lasting at least 60 minutes; and
8. consent to participate in the study.

Exclusion Criteria:

1. prior neurological or psychiatric disorders;
2. severe spasticity (Modified Ashworth Scale >3) over hemiplegic upper extremity;
3. a history of recent Botox injections or acupuncture to the hemiplegic upper extremity within the past three months;
4. use of central nervous system-active medicine;
5. any contraindication to TMS, according to the guideline of the Safety of TMS Consensus group, such as the risk of epilepsy, metal implants, and pregnancy;
6. the presence of unilateral neglect as screened by the Behavioural Inattention Test (CBIT-HK); and
7. participation in another clinical study elsewhere during recruitment. Informed written consent will be obtained from all patients prior to data collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment (FMA) | Baseline
  A stroke-specific, performance-based impairment index
Fugl-Meyer assessment (FMA) | 1 day
  A stroke-specific, performance-based impairment index
Fugl-Meyer assessment (FMA) | 2 weeks
  A stroke-specific, performance-based impairment index
Fugl-Meyer assessment (FMA) | 1-month after the completion of the intervention
  A stroke-specific, performance-based impairment index
Action Research Arm Test (ARAT) | Baseline (immediately before the first session)
  A measure of upper extremity performance (coordination, dexterity and functioning) in stroke recovery
Action Research Arm Test (ARAT) | 1 day
  A measure of upper extremity performance (coordination, dexterity and functioning) in stroke recovery
Action Research Arm Test (ARAT) | 2 weeks
  A measure of upper extremity performance (coordination, dexterity and functioning) in stroke recovery
Action Research Arm Test (ARAT) | 1-month after the completion of the intervention
  A measure of upper extremity performance (coordination, dexterity and functioning) in stroke recovery

SECONDARY OUTCOMES:
EEG rhythm power | Baseline (immediately before the first session)
  Rhythm power desynchronization/synchronization in response to mirror visual feedback
EEG rhythm power | 1 day
  Rhythm power desynchronization/synchronization in response to mirror visual feedback
EEG rhythm power | 2 weeks
  Rhythm power desynchronization/synchronization in response to mirror visual feedback
EEG rhythm power | 1-month after the completion of the intervention
  Rhythm power desynchronization/synchronization in response to mirror visual feedback
Motor-evoked Potential (MEP) | Baseline (immediately before the first session)
  Electrical potential recorded over a hand muscle, evoked by stimulating the primary motor cortex.
Motor-evoked Potential (MEP) | 1 day
  Electrical potential recorded over a hand muscle, evoked by stimulating the primary motor cortex.
Motor-evoked Potential (MEP) | 2 weeks
  Electrical potential recorded over a hand muscle, evoked by stimulating the primary motor cortex.
Motor-evoked Potential (MEP) | 1-month after the completion of the intervention
  Electrical potential recorded over a hand muscle, evoked by stimulating the primary motor cortex
Cortical silent period | Baseline (immediately before the first session)
  The cortical silent period (cSP) refers to an interruption of voluntary muscle activities during contraction by stimulating the contralateral primary motor cortex.
Cortical silent period | 1 day
  The cortical silent period (cSP) refers to an interruption of voluntary muscle activities during contraction by stimulating the contralateral primary motor cortex.
Cortical silent period | 2 weeks
  The cortical silent period (cSP) refers to an interruption of voluntary muscle activities during contraction by stimulating the contralateral primary motor cortex.
Cortical silent period | 1-month after the completion of the intervention
  The cortical silent period (cSP) refers to an interruption of voluntary muscle activities during contraction by stimulating the contralateral primary motor cortex.
Ipsilateral silent period | Baseline (immediately before the first session)
  Ipsilateral silent period (iSP) is an interruption of ongoing muscle activities caused by stimulating ipsilateral primary motor cortex.
Ipsilateral silent period | 1 day
  Ipsilateral silent period (iSP) is an interruption of ongoing muscle activities caused by stimulating ipsilateral primary motor cortex.
Ipsilateral silent period | 2 weeks
  Ipsilateral silent period (iSP) is an interruption of ongoing muscle activities caused by stimulating ipsilateral primary motor cortex.
Ipsilateral silent period | 1-month after the completion of the intervention
  Ipsilateral silent period (iSP) is an interruption of ongoing muscle activities caused by stimulating ipsilateral primary motor cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Nai Kuen FONG, PHD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Kenneth FONG, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided